CLINICAL TRIAL: NCT01899521
Title: Alcohol Abuse, Oxidative Stress, and Zinc Deficiency in Lung Disease
Brief Title: Examination of Zinc, S-adenosylmethionine, and Combination Therapy Versus Placebo in Alcoholics
Acronym: ExZACTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PULM-038-12S; IRB00060773 (Other: Emory IRB); IK2CX000643 (NIH)
Record Dates: First submitted 2013-06-27; First posted 2013-07-15 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Alcoholism
Keywords: alcoholism; lung health; pulmonary; macrophage; zinc; SAMe; S-adenosylmethionine; alveolar
MeSH Terms: conditions — Alcoholism | interventions — Bronchoscopy; Zinc Sulfate; S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo zinc and placebo SAMe (Placebo Comparator): Placebo tablet of zinc sulfate once daily and placebo tablet of s-adenosylmethionine twice daily
  Interventions: Procedure: Bronchoscopy
- Active zinc and placebo SAMe (Active Comparator): Zinc sulfate 220 mg once daily and placebo tablet of s-adenosylmethionine twice daily
  Interventions: Procedure: Bronchoscopy; Dietary Supplement: Zinc sulfate 220 mg once daily
- Placebo zinc and active SAMe (Active Comparator): Placebo tablet of zinc sulfate once daily and s-adenosylmethionine 400 mg twice daily
  Interventions: Procedure: Bronchoscopy; Dietary Supplement: S-adenosylmethionine 400 mg twice daily
- Active zinc and active SAMe (Active Comparator): Zinc sulfate 220 mg once daily and s-adenosylmethionine 400 mg twice daily
  Interventions: Procedure: Bronchoscopy; Dietary Supplement: Zinc sulfate 220 mg once daily; Dietary Supplement: S-adenosylmethionine 400 mg twice daily

INTERVENTIONS:
Procedure: Bronchoscopy — Involves flexible fiberoptic bronchoscopy with standardized bronchoalveolar lavage (BAL) technique (isotonic saline in a sub-segment of the right middle lobe or lingula) using standard conscious sedation techniques.
Dietary Supplement: Zinc sulfate 220 mg once daily
  Arms: Active zinc and active SAMe; Active zinc and placebo SAMe
Dietary Supplement: S-adenosylmethionine 400 mg twice daily
  Other Names: SAMe
  Arms: Active zinc and active SAMe; Placebo zinc and active SAMe

SUMMARY:
This is a randomized, placebo controlled trial of dietary zinc and S-adenosylmethionine (SAMe) in otherwise healthy alcoholic US Veterans. The primary goal is to determine if either dietary zinc or S-adenosylmethionine (SAMe) can augment lung immune defenses in alcoholics and thereby decrease the risk of lung injury and infection.

DETAILED DESCRIPTION:
Alcohol abuse is a major burden on society and even more of a problem in the Veteran population. Chronic alcohol ingestion can have serious health consequences including pneumonia and acute lung injury, which can occur suddenly and without warning even in physically fit individuals without apparent signs of alcohol dependence. Therefore, it is vital for the health of our Veterans and indeed the entire population to identify effective treatments that can limit or even prevent these devastating consequences. The primary goal of this clinical research project is to determine if dietary zinc or supplements of the antioxidant S-adenosylmethionine (SAMe) can augment lung immune defenses in otherwise healthy alcoholics and thereby decrease the risk of lung injury and infection. There is already strong evidence from the investigators' experimental animal model that moderate daily alcohol ingestion for as little as six weeks causes oxidative stress and zinc deficiency in the lung. These derangements result insult in dysfunction of the alveolar macrophage, which is the resident immune cell, and predisposes animals to the development of pneumonia. Importantly, in this same animal model, the investigators found that adding either zinc or antioxidants to the diet prevents these problems and preserves lung health even during daily alcohol ingestion.

This project will translate basic findings in the animal model to the clinical setting and determine whether or not zinc or SAMe supplements are effective in humans who pathologically consume alcohol. This project will enroll Veterans seen at the Atlanta Veterans Hospital in the Substance Abuse Treatment Program (SATP). Participants will be evaluated by undergoing a procedure to obtain samples of fluid from their lungs, measure zinc levels, redox potential, and assess how well their alveolar macrophages respond to bacteria (by determining phagocytic capacity). After completion of the initial evaluation, the participants will be randomized to receive standard treatment (placebo), zinc supplements, dietary SAMe, or the combination of zinc and SAMe for 14 days. All subjects will be evaluated for two weeks as they undergo treatment. At the end of this two week period, measurements of lung zinc, redox potential and macrophage function will be repeated and compared between the two groups. The hypothesis is that both dietary zinc and SAM supplements will improve the immune function of the alveolar macrophage.

If this project is successful, it will lead to larger clinical trials to determine if either dietary zinc and/or SAMe supplements can be effective even in the acute clinical setting and improve outcomes in alcoholics who develop pneumonia or acute lung injury. Overall, both zinc and SAMe supplements are safe and inexpensive to provide, allowing these potential treatments to be easily implemented in the Veteran population as well as society in general. Given the significant burden of unhealthy alcohol use, the investigators need ways to limit the physical consequences of alcohol abuse while the investigators continue the efforts at public education and addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Active alcohol use disorder

Exclusion Criteria:

* Any active and uncontrolled medical problem(s)
* Known zinc deficiency
* Primary substance of abuse something other than alcohol
* Current abnormal chest x-ray
* HIV-positive
* Any disorder of blood coagulation
* Currently on medical treatment with anti-coagulants, including:

  * warfarin
  * heparin
  * direct thrombin inhibitors
  * anti-platelet agents (other than Aspirin)
* Daily use of vitamins or other nutritional supplements (unless taking as treatment for alcohol use disorder)
* Renal impairment (GFR < 60)
* Active bipolar disorder
* Active Parkinson's disease
* Current pregnancy
* Contraindication to treatment with zinc or S-adenosylmethionine
* Inability to give informed consent (i.e., limited cognitive capacity)
* Non-English speaking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Mehta, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants are enrolled when they sign consent, however, only get randomized after completing first bronchoscopy procedure. Therefore, there were some participants who enrolled but never completed the procedure in order to be randomized into a group. This is the reason for the discrepancy in numbers.
Groups:
- Active Zinc and Placebo SAMe: Zinc sulfate 220 mg once daily and placebo tablet of s-adenosylmethionine twice daily
  Bronchoscopy: Involves flexible fiberoptic bronchoscopy with standardized bronchoalveolar lavage (BAL) technique (isotonic saline in a sub-segment of the right middle lobe or lingula) using standard conscious sedation techniques.
  Zinc sulfate 220 mg once daily
- Placebo Zinc and Active SAMe: Placebo tablet of zinc sulfate once daily and s-adenosylmethionine 400 mg twice daily
  Bronchoscopy: Involves flexible fiberoptic bronchoscopy with standardized bronchoalveolar lavage (BAL) technique (isotonic saline in a sub-segment of the right middle lobe or lingula) using standard conscious sedation techniques.
  S-adenosylmethionine 400 mg twice daily
- Active Zinc and Active SAMe: Zinc sulfate 220 mg once daily and s-adenosylmethionine 400 mg twice daily
  Bronchoscopy: Involves flexible fiberoptic bronchoscopy with standardized bronchoalveolar lavage (BAL) technique (isotonic saline in a sub-segment of the right middle lobe or lingula) using standard conscious sedation techniques.
  Zinc sulfate 220 mg once daily
  S-adenosylmethionine 400 mg twice daily
Period: Overall Study
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe
Started | 23 | 25 | 25 | 22
Completed | 18 | 24 | 24 | 20
Not Completed | 5 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe | Total
Number analyzed (Participants) | 23 | 25 | 25 | 22 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 25 | 22 | 95
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 46 [28 to 60] | 47 [28 to 58] | 47 [29 to 60] | 51 [27 to 60] | 48 [27 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 4 | 15
  Male | 21 | 21 | 20 | 18 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 22 | 25 | 24 | 21 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 20 | 21 | 19 | 77
  White | 4 | 2 | 2 | 2 | 10
  More than one race | 2 | 3 | 2 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 25 | 22 | 95
Smoking Status [Count of Participants; unit: Participants]
  Smoker | 14 | 15 | 15 | 14 | 58
  Non-smoker | 9 | 10 | 10 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint
Description: Improvement in alveolar macrophage phagocytic index. Phagocytic index will be measured before and after treatment phase. Phagocytic index is calculated using isolated alveolar macrophages from the bronchoscopy procedure such that phagocytic index = (total number of engulfed cells/total number of counted macrophages) x (number of macrophages containing engulfed cells/total number of counted macrophages) x 100.
Time Frame: Initial bronchoscopy to second bronchoscopy (Initial bronchoscopy performed prior to treatment and second bronchoscopy done 2-3 weeks after starting treatment)
Measure: Mean (Standard Deviation); unit: Phagocytic Index (PI)
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe
Number analyzed (Participants) | 18 | 24 | 24 | 20
Phagocytic Index (PI)
  Pre-treatment PI | 13518 (11677) | 15892 (18961) | 10849 (11087) | 15530 (17627)
  Post-treatment PI | 16704 (15412) | 23850 (47703) | 10734 (9709) | 13955 (14511)

2. Secondary Outcome: Secondary Endpoint
Description: Improvement in alveolar macrophage intracellular zinc. Intracellular zinc will be measured before and after treatment phase using isolated alveolar macrophages. The units of measure are relative fluorescence units/cell (RFU/cell) and measured using confocal microscopy techniques.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: RFU/cell
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe
Number analyzed (Participants) | 18 | 24 | 24 | 20
RFU/cell
  Pre-treatment Intracellular Zinc | 2816 (2149) | 3410 (2655) | 3883 (2723) | 4174 (3386)
  Post-treatment Intracellular Zinc | 2710 (1980) | 3510 (2590) | 4327 (3092) | 3103 (2823)

3. Other Pre Specified Outcome: Secondary Endpoint
Description: Improvement in redox potential in the alveolar space. Redox potential will be measured before and after treatment phase using lavage fluid and blood plasma.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: GSSG percentage (measure of oxidation)
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe
Number analyzed (Participants) | 18 | 24 | 24 | 20
GSSG percentage (measure of oxidation)
  Pre-treatment GSSG | 33.0 (30.5) | 28.0 (29.2) | 21.6 (25.3) | 28.5 (30.6)
  Post-treatment GSSG | 28.9 (29.2) | 19.7 (23.8) | 20.5 (26.8) | 33.5 (35.2)

4. Other Pre Specified Outcome: Secondary Endpoint
Description: Improvement in alveolar macrophage granulocyte macrophage - colony stimulating factor (GM-CSF) receptor expression. GM-CSF receptor expression will be measured before and after treatment phase using isolated alveolar macrophages. The units of measure are relative fluorescence units/cell (RFU/cell) and measured using confocal microscopy techniques. Both alpha- and beta-subunits of the receptor will be measured.
Time Frame: as for outcome 1
Population: The cells were not stained appropriately, so this secondary measure could not be completed because the results were not analyzable.
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: Secondary Endpoint
Description: Improvement in serum zinc level. Serum zinc will be measured before and after treatment phase by collecting blood plasma. The units of measure are mcg/dl.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/dl
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe
Number analyzed (Participants) | 18 | 24 | 24 | 20
mcg/dl
  Pre-treatment Serum Zinc | 79.5 (18.5) | 76.9 (12.0) | 78.5 (12.1) | 75.0 (11.0)
  Post-treatment Serum Zinc | 71.2 (9.7) | 95.6 (36.3) | 80.1 (14.9) | 92.0 (34.8)

ADVERSE EVENTS:
Time Frame: Up to one month following the final bronchoscopy procedure, a total of about two months. Subjects were assessed while they were enrolled and taking study medications and completed all study procedures after the second bronchoscopy. They were contacted from day following procedure up to a total 4 weeks after the final procedure date to assess for any additional adverse events. The total time period is about two months, including time during the study and after the final bronchoscopy procedure.
Arm/Group | Placebo Zinc and Placebo SAMe | Active Zinc and Placebo SAMe | Placebo Zinc and Active SAMe | Active Zinc and Active SAMe
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25 | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/25 | 1/25 | 0/22
Other Adverse Events (participants affected / at risk) | 17/23 | 21/25 | 16/25 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Zinc and Placebo SAMe (N=23) | Active Zinc and Placebo SAMe (N=25) | Placebo Zinc and Active SAMe (N=25) | Active Zinc and Active SAMe (N=22)
Subarachnoid hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Zinc and Placebo SAMe (N=23) | Active Zinc and Placebo SAMe (N=25) | Placebo Zinc and Active SAMe (N=25) | Active Zinc and Active SAMe (N=22)
GI upset (Gastrointestinal disorders) | 5 (5) | 8 (10) | 7 (8) | 11 (16) — May be diarrhea, upset stomach, flatulence
Procedure-related (Injury, poisoning and procedural complications) | 8 (13) | 9 (10) | 8 (9) | 6 (6) — Includes sore throat, chest soreness, cough
Other (Investigations) | 6 | 9 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT01899521/Prot_SAP_000.pdf